CLINICAL TRIAL: NCT06678802
Title: ROLE OF CIRCULATING SMALL NUCLEOLAR RNA SNORD3A IN ISCHEMIC HEART DISEASE AND HEART FAILURE
Brief Title: SNORD3A IN ISCHEMIC HEART DISEASE AND HEART FAILURE
Acronym: SENSITISE
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giovanni Esposito, Professor, Director, Federico II University
Other Study IDs: 273/2023
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-03

CONDITIONS: Ischemic Heart Disease; Heart Failure
MeSH Terms: conditions — Myocardial Ischemia; Heart Failure | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1 - Chronic ischemic heart disease
  Interventions: Other: Blood sampling
- 2 - Acute coronary syndromes
  Interventions: Other: Blood sampling
- 3 - Healthy volunteers
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — blood sampling from peripheral vein

SUMMARY:
This is a prospective, non-randomized, single center, open label clinical study enrolling patients affected by 1) chronic ischemic heart disease with evidence or suspect significant myocardial ischemia (group 1, CCS) or 2) acute coronary syndromes (group 2, ACS), both undergoing coronary angiography and eventually coronary revascularization at the Department of Scienze Cardiovascolari, Diagnostica per Immagini ed Emergenze Cardiovascolari of Federico II University Hospital, Naples, Italy. Age and sex-matched healthy volunteers without known ischemic heart disease (group 3, Ctr) will also be included as a control group. At enrollment (time 0), and after 48 hours (time 48 h), 1 month (time 1mo) and 6 month-follow-up visits (time 6 mo), clinical evaluation, ECG, trans-thoracic echocardiography and blood sampling will be performed, to isolate peripheral blood mononuclear cells (PBMC) and perform standard blood tests. The enrolment phase will last 24 months, and will likely involve 450 patients distributed as follows, according to the number of patients annually referring to our University

Hospital:

1. Group 1, n= 200 patients with chronic ischemic heart disease undergoing coronary angiography and eventually coronary revascularization;
2. Group 2, n= 200 patients with ACS undergoing coronary angiography and eventually coronary revascularization ;
3. Group 3, n= 50, healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

History (> 6 months) of ischemic heart disease (prior myocardial infarction, prior percutaneous coronary intervention, prior surgical revascularization) and clinical or imaging evidence of chronic moderate or severe myocardial ischemia

Group 2:

Patients with acute coronary syndromes at presentation including ST-elevation myocardial infarction, Non-ST elevation myocardial infarction, and unstable angina.

Group 3:

Healthy volunteers with no prior history of ischemic heart disease or clinical/imaging evidence of myocardial ischemia.

Exclusion Criteria:

Patients unwilling to provide informed consent to participate to the study

* Concomitant primary cardiomyopathies or hemodynamically significant heart valve disease
* Treatment with cancer or antibiotic therapies affecting ribosomal structure or function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective, non-randomized, single center, open label clinical study enrolling patients affected by 1) chronic ischemic heart disease with evidence or suspect significant myocardial ischemia (group 1, CCS) or 2) acute coronary syndromes (group 2, ACS), both undergoing coronary angiography and eventually coronary revascularization at the Department of Scienze Cardiovascolari, Diagnostica per Immagini ed Emergenze Cardiovascolari of Federico II University Hospital, Naples, Italy. Age and sex-matched healthy volunteers without known ischemic heart disease (group 3, Ctr) will also be included as a control group. At enrollment (time 0), and after 48 hours (time 48 h), 1 month (time 1mo) and 6 month-follow-up visits (time 6 mo), clinical evaluation, ECG, trans-thoracic echocardiography and blood sampling will be performed, to isolate peripheral blood mononuclear cells (PBMC) and perform standard blood tests.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | 0, 1 month, 6 months
NT-pro-BNP levels | 0, 1 month, 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University Hospital, Naples, Italy

IPD SHARING:
Plan to Share IPD: No